CLINICAL TRIAL: NCT05470725
Title: A Phase 1, Open-Label, Single-Dose, Parallel-Group Study to Evaluate the Pharmacokinetics of CIN-107 in Subjects With Varying Degrees of Renal Function
Brief Title: Study to Evaluate the Pharmacokinetics of CIN-107 in Subjects With Varying Degrees of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIN-107-113
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control (normal renal function or mild renal impairment) (Experimental): Estimated glomerular filtration rate (eGFR) ≥60 mL/min
  Interventions: Drug: CIN-107
- Moderate to severe renal impairment (Experimental): eGFR 15 to 59 mL/min
  Interventions: Drug: CIN-107
- Kidney failure (Experimental): eGFR <15 mL/min, including:
  * Subjects not on dialysis; and
  * Subjects on dialysis, with study drug administration on a non-dialysis day
  Interventions: Drug: CIN-107

INTERVENTIONS:
Drug: CIN-107 — A single 10 mg CIN-107 oral dose (2 X 5 mg tablets).
  Other Names: baxdrostat

SUMMARY:
This is a Phase 1, open-label, parallel-group study in subjects with varying degrees of renal function to assess the safety, tolerability, and Pharmacokinetics of a single 10 mg oral dose of CIN-107.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in stable health based on medical and psychiatric history, physical examination, ECG, vital signs (seated and orthostatic), and routine laboratory tests (chemistry, hematology, coagulation, and urinalysis); Note: Underlying medical conditions consistent with the population under study are acceptable if the subject's condition is considered stable by the Investigator. For renally impaired subjects, their renal status must be stable for a minimum of 3 months prior to screening.
* Does not use nicotine-containing products at all or smokes <10 cigarettes/day (approximately <half pack/day);
* Body mass index (BMI) between 18 and 40 kg/m2, inclusive;

Exclusion Criteria:

* Active participation in another experimental therapy study of a small molecule other than CIN-107 within 30 days prior to Day 1 or 5 half-lives, whichever is longer; or received a large molecule within 90 days prior to Day 1 or 5 half-lives, whichever is longer;
* History of prior organ transplant or planned transplant within 6 months of screening;
* Personal or family history of long QT syndrome, torsades de pointes, or other complex ventricular arrhythmias, or family history of sudden death;
* History of, or current, clinically significant arrhythmias as judged by the Investigator, including ventricular tachycardia, ventricular fibrillation, chronic persistent atrial fibrillation, sinus node dysfunction, or clinically significant heart block. Subjects with minor forms of ectopy (eg, premature atrial contractions) are not necessarily excluded;
* Prolonged QTcF (>450 msec for males or >470 msec for females) based on the average of triplicate ECGs;
* Evidence of any of the following clinical measurements:

  1. Seated systolic BP >160 mmHg and/or diastolic BP >100 mmHg, or systolic BP <90 mmHg and/or diastolic BP <50 mmHg;
  2. Resting heart rate >100 beats per minute (bpm) or <50 bpm;
  3. Oral temperature >37.6°C (>99.68°F);
  4. Respiration rate 20 breaths/minute;
  5. Postural tachycardia (ie, an increase in heart rate >30 bpm upon standing from a seated position);
  6. Orthostatic hypotension (ie, a fall in systolic BP ≥20 mmHg or diastolic BP ≥10 mmHg upon standing from a seated position);
  7. Clinically significant abnormal serum potassium >upper limit of normal of the reference range (ULN);
  8. Clinically significant abnormal serum sodium 1.5 x ULN;
  9. Aspartate aminotransferase or alanine aminotransferase values >1.5 x ULN
  10. Total bilirubin >2 x ULN, unless due to Gilbert's syndrome;
  11. Positive test for HIV antibody, hepatitis C virus (HCV) RNA, hepatitis B surface antigen (HBsAg), or SARS-CoV-2 RNA; or
* History of porphyria, myopathy, or active liver disease;
* Inadequate venous access;
* Current treatment with weight loss medication or prior weight loss surgery (eg, gastric bypass surgery);
* Use of a strong inducer of CYP3A4 within 28 days prior to the dose of study drug;
* Corticosteroid use (systemic or extensive topical use) within 3 months prior to study drug dosing;
* Positive drug or alcohol test result without medical explanation or a history of alcoholism or drug abuse within 2 years prior to study drug dosing as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition;
* Typical consumption of ≥14 alcoholic drinks weekly;
* Surgical procedures within 4 weeks prior to study drug dosing or planned elective surgery during the study period;
* Any clinically significant illness within 4 weeks prior to study drug dosing, unless deemed not clinically significant by the Investigator;
* Pregnant, breastfeeding, or planning to become pregnant during the study;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to Day 8
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data, as the data permit.
Time to maximum plasma concentration (Tmax) | up to Day 8
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data, as the data permit.
Area under the curve from time 0 to the time of last quantifiable plasma concentration (AUC[0-last]) | up to Day 8
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data, as the data permit.
Area under the curve from time 0 to infinity (AUC[0-inf]) | up to Day 8
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data, as the data permit.
Percent of AUC extrapolated | up to Day 8
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data, as the data permit.
Terminal phase elimination half-life | up to Day 8
  This PK parameter will be determined for CIN-107, its primary metabolite (CIN-107-M), and any other measured metabolites using plasma concentration data, as the data permit.
Apparent plasma clearance (CL/F) | up to Day 8
  This PK parameter will be determined for CIN-107 using plasma concentration data.
Apparent volume of distribution | up to Day 8
  This PK parameter will be determined for CIN-107 using plasma concentration data.
The cumulative amount of CIN-107 and CIN-107-M excreted in the urine (Ae) | up to Day 8
  This PK parameter will be calculated using the urine concentrations of CIN-107 and its primary metabolite (CIN-107-M)
Renal clearance (CLR) of CIN-107 and CIN-107-M of CIN-107 and CIN-107-M | up to Day 8
  Calculated as Ae/AUC. This PK parameter will be calculated using the urine concentrations of CIN-107 and its primary metabolite (CIN-107-M)
The fraction of the dose excreted renally | up to Day 8
  This PK parameter will be calculated using the urine concentrations of CIN-107
Number of patients experiencing adverse events (AEs) | up to Day 11
Number of patients experiencing adverse drug reactions | up to Day 11
Number of patients experiencing serious adverse events (SAEs) | up to Day 11

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Trials, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=CIN-107-113&attachmentIdentifier=470157a5-c75d-4658-984f-d465ba903b3e&fileName=cin-107-113-report-synopsis_Redacted.pdf&versionIdentifier=